CLINICAL TRIAL: NCT04191525
Title: A 12 Week, Randomized, Double-blind, Placebo-controlled, Phase II Trial to Evaluate the Efficacy and Safety of the Treatment With BPL-1 in Adult Patients With Type 2 Diabetes Mellitus With Different Course of Disease and Treatment
Brief Title: Phase II Clinical Trial to Evaluate the Efficacy and Safety of the Treatment With BPL-1 in Adult Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mónica Marazuela Azpíroz (Other)
Collaborators: Alba Garcimartín Álvarez (Unknown); Carolina Knott Torcal (Unknown); Nerea Aguirre Moreno (Unknown); Miguel Antonio Sampedro Núñez (Unknown); María Caldas (Unknown); Belén Ruiz-Rosso (Unknown); Ana María Ramos Levi (Unknown)
Responsible Party: Sponsor-Investigator, Mónica Marazuela Azpíroz, Head of Endocrinology and Nutrition, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROBIDEM
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Microbiote; Cardiovascular Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Single-centre, randomized, double-blind clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPL-1 Probiotic capsules (Experimental): BPL-1 Probiotic 1 capsule/day
  Interventions: Dietary Supplement: BPL-1 Probiotic capsules
- Placebo (Placebo Comparator): 1 capsule/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BPL-1 Probiotic capsules — BPL-1 Probiotic 1 capsule/day
  Arms: BPL-1 Probiotic capsules
Dietary Supplement: Placebo — Placebo masked with the same presentation as the experimental product 1 capsule/day
  Arms: Placebo

SUMMARY:
Diabetes Mellitus type 2 (T2DM) is a chronic and progressive disease, characterized mainly by hyperglycemia. Metabolic imbalance causes an increased risk of microvascular and macrovascular complications associated with the increased prevalence of cardiovascular disease (CVD) in diabetics.

Although genetic predisposition determines individual susceptibility to T2DM, external factors such as an unhealthy diet and a sedentary lifestyle condition the onset of the disease.

Since T2DM is a multifactorial disease, many authors have studied the possible role of the microbiota and its alterations in the pathophysiology of the disease. There is evidence that in T2DM there are alterations in the proportion of Firmicutes, Bacteroidetes and Proteobacteria, and a smaller amount of bifidobacteria with anti-inflammatory properties.

Probiotics are living microorganisms present in food that, if consumed in sufficient quantities, can improve health. In general, probiotics protect the patient through immunomodulation, protecting him from infections, increasing the activation of mononuclear cells and lymphocytes.

The investigational product is a supplement to the probiotic Bifidobacterium animalis subsp. lactis (BPL-1) CECT 8145. There are numerous studies carried out on different strains of GLP-1 that demonstrate its safety. Many of them are commonly used in the food industry, not only because of their proven safety, but also because of their viability until consumption.

This clinical trial is proposed as an interdisciplinary study that can contribute to the characterization of the efficacy of treatment with probiotics in patients with T2DM of different stages of evolution, without and with hepatic involvement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18-75 (inclusive)
* BMI ≥ 27
* Glycated hemoglobin > 5,6 and/or fasting glucose > 100 mg/dl and/or being on active treatment with at least one antidiabetic medication
* Subjects must be able to provide written informed consent
* Females of childbearing potential must have a previous negative pregnancy test and must agree to use adequate contraception during their participation in the study

Exclusion Criteria:

* Crohn's disease, liver cirrhosis, human immunodeficiency virus (HIV) or any other active systemic bacterial, viral or fungal infections
* BMI > 42
* Severe hypoglycemias within 3 months prior to the start date of the study
* Abnormal glycated hemoglobin measurements (over 8%) prior to the start date of the study
* Prescription of a new antidiabetic medication in the last 6 months
* Celiac disease or any other food intolerances
* Use of antibiotics, probiotics and/or prebiotics within 2 weeks prior to the start date of the study
* Chronic liver disease with a C Child-Plug score, chronic kidney disease with creatinine clearance < 50 ml/min as well as any other clinically significant conditions including pulmonary, neurological and cardiovascular diseases according to the investigators medical opinion
* Patients with history or presence of malignancy who have been treated with systemic antineoplastic therapy within 6 months prior to the start date of the study
* Pregnancy and breastfeeding
* Not being able to provide written informed consent to participate in the study or to cooperate and comply with the study procedures for any other reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | 12 weeks
  Fasting glucose
Glycated haemoglobin | 12 weeks
  Glycated haemoglobin
Insulin | 12 weeks
  Insulin
HOMA-IR | 12 weeks
  HOMA-IR

SECONDARY OUTCOMES:
Total cholesterol | 12 weeks
  Total cholesterol
HDL-cholesterol | 12 weeks
  HDL-cholesterol
LDL-cholesterol | 12 weeks
  LDL-cholesterol
Triglycerides | 12 weeks
  Triglycerides
Body Mass Index (BMI) | 12 weeks
  Body Mass Index (BMI)
Body Fat Percentage (%BF) | 12 weeks
  Body Fat Percentage (%BF)
Blood pressure | 12 weeks
  Blood pressure
Waist perimeter | 12 weeks
  Waist perimeter

OTHER OUTCOMES:
Mediterranean diet adherence score | 12 weeks
  Mediterranean diet adherence score

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Marazuela Azpíroz, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de La princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No